CLINICAL TRIAL: NCT06258499
Title: A Multicenter, Randomized, Controlled, Blinded Study of the Safety and Efficacy of Bone Healing Accelerant Versus Autologous Bone Grafting in Subjects Undergoing Hindfoot or Ankle Arthrodesis and Who Require Supplementary Grafting
Brief Title: Bone Healing Accelerant (BHA) Versus Autologous Bone Grafting (ABG) for Hindfoot or Ankle Arthrodesis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: study never started and is on hold until further notice
Sponsor: Carmell Therapeutics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAR-BHA- U22
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Foot Deformities
MeSH Terms: conditions — Foot Deformities | interventions — Butylated Hydroxyanisole

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- BHA (Experimental): Subjects treated with BHA + standard of care
  Interventions: Combination Product: BHA
- Control (No Intervention): Subjects treated as per standard of care

INTERVENTIONS:
Combination Product: BHA — BHA active ingredients include a blood-derived component and beta-tricalcium phosphate. It is manually placed into the joint fusion space during fusion surgery.
  Arms: BHA

SUMMARY:
This study is being conducted to demonstrate the safety and effectiveness of Bone Healing Accelerant (BHA) product when applied to the joint space of the ankle of hindfoot (the section of the foot immediately below the ankle joint) during fusion surgery. It is hypothesized that by 6 months, the number of subjects with successful bone fusion will be greater in the BHA-treated group compared to subjects treated with standard of care alone.

ELIGIBILITY:
Inclusion Criteria:

* Patient has pain with weight-bearing in the joint(s) below that, in the opinion of the Investigator, warrants arthrodesis:

  1. Tibiotalar (ankle)
  2. Talocalcaneal (subtalar)
  3. Talonavicular
  4. Calcaneocuboid
  5. Double hindfoot (e.g., talonavicular and talocalcaneal joints)
  6. Triple hindfoot (subtalar, talonavicular and calcaneocuboid joints
* Joint space(s) can, in the opinion of the Investigator, be adequately filled with no more than 9 cc of graft material (BHA or ABG)
* Each fused joint can be adequately compressed and rigidly stabilized with plates, screws, staples or a combination thereof. External fixation, percutaneous Kirschner wires or intramedullary rods may not be used.
* Patient is willing and able to comply with all study requirements including all postoperative clinical and radiographic evaluations.
* If patient is a woman of childbearing bearing potential (not post-menopausal for 12 months or surgically sterile), patient has a urine pregnancy test with a negative result at screening and on the day of surgery, prior to the procedure. These trial participants must commit to adequate birth control through the 52-week follow-up

Exclusion Criteria:

* Skeletally immature patients (i.e., radiographic evidence of open physes), regardless of age
* Bone deficit, defect or void requiring a structural graft
* Condition requiring intramedullary nailing or external fixation for the arthrodesis
* Condition requiring osteotomy or fusion of any midfoot joints.
* Prior arthroplasty, arthrodesis, major surgical repair or reconstruction of the index ankle or hindfoot joints.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Successful Radiographic Fusion | 24 weeks
  Greater than or equal to 50% bone bridging across joint space for the full complement of joints fused as determined by CT in the absence of secondary surgical or nonsurgical interventions intended to promote fusion.